CLINICAL TRIAL: NCT03440645
Title: Cardiovascular Screening for Family Members of People With Acute Coronary Disease: A Patient-Initiated and Family-Oriented Strategy
Brief Title: Cardiovascular Screening for Family Members of People With Acute Coronary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Michael Goldfarb, Clinician-Investigator, Lady Davis Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pending
Record Dates: First submitted 2018-01-04; First posted 2018-02-22 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family or Household Members (Experimental)
  Interventions: Other: Family-oriented primary cardiovascular prevention

INTERVENTIONS:
Other: Family-oriented primary cardiovascular prevention — An initial screening visit including a targeted history, physical exam, and investigations as per the Canadian Cardiovascular Society's recommendations for cardiovascular primary prevention. Counselling and informational handouts on improved cardiovascular risk factor and lifestyle habits. All family and household members, as well as the cardiovascular disease proband, are encouraged to attend and participate in all healthcare visits.

SUMMARY:
Over a 12-month period, patients admitted with acute coronary disease to the cardiovascular care unit at the Jewish General Hospital (JGH), an academic tertiary care referral center in Montreal, Quebec, will be approached to refer first-degree relatives and/or household members age 18 years or older to an outpatient cardiovascular (CV) risk factor screening and treatment program. Relatives and household members will undergo a focused history, physical, and CV risk factor assessment and will receive evidence-based guideline-recommended treatment as indicated. Participants will be referred to nutritionists, smoking cessation programs, and to other allied healthcare professionals as needed. A follow-up visit at 6-months will assess treatment adherence and improvement in CV risk factors. All family and/or household members including the index patient will be encouraged to attend all healthcare visits together.

The effectiveness of the screening strategy will be measured by the total number of participants identified as intermediate or high modified Framingham 10-year risk of cardiovascular disease. The effectiveness of the primary prevention intervention will be measured by the change in percentage of the mean modified Framingham 10-year risk score for participants between the initial visit and 6-month follow-up. The value of the referral, screening, and treatment program, as well as participant engagement and satisfaction will also be systematically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≤70 years old admitted with an initial diagnosis of an acute coronary event (such as acute coronary syndrome or myocardial infarction)
* At least 1 first-degree family or household member age ≥ 18 years old

Exclusion Criteria

* No eligible family or household members
* Inability to contact family or household members
* Distance to study centre too far as determined by the patient
* Family or household members who have been screened for CV disease in the previous 2 years.
* Family or household members with known coronary disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Change in mean modified Framingham cardiovascular risk score from the initial visit to the 6 month follow-up visit | 6 months
  The change in percentage of the mean modified Framingham cardiovascular risk score for family and household members between the initial visit and the 6-month follow-up visit

SECONDARY OUTCOMES:
Effectiveness of the screening strategy | 12 months of study recruitment
  Total number of participants identified at intermediate or high risk on the modified Framingham CV risk score

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldfarb, MD, Principal Investigator — Lady Davis Institute for Medical Research
Locations (1):
- Jewish General Hospital / Lady Davis Institute, Montreal, Quebec, Canada

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT03440645/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT03440645/ICF_001.pdf